CLINICAL TRIAL: NCT04965103
Title: Graft Reconstruction for Irreparable Rotator Cuff Tears: Superior Capsule Reconstruction or Tendon Repair With Graft Interposition
Brief Title: Superior Capsule vs Bridging Study
Acronym: SCR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Collaborators: Worker's Compensation Board of Alberta (funding) (Unknown); Canadian Orthopaedic Foundation (funding) (Unknown); Arthroscopy Association of North America (funding) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REB15-1787
Record Dates: First submitted 2021-06-21; First posted 2021-07-16 (Actual); Last update posted 2021-07-16 (Actual); Status verified 2021-06

CONDITIONS: Rotator Cuff Tears
Keywords: irreparable
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participant and research assistant collecting outcomes were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bridging (Active Comparator): Tendon repair with graft interposition
  Interventions: Procedure: Bridging
- SCR (Experimental): Superior Capsule reconstruction
  Interventions: Procedure: SCR

INTERVENTIONS:
Procedure: SCR — Superior Capsule reconstruction
  Arms: SCR
Procedure: Bridging — Tendon repair with graft interposition
  Arms: Bridging

SUMMARY:
Randomized controlled trial examining superior capsule reconstruction versus tendon repair with graft interposition in "irreparable" rotator cuff tears.

DETAILED DESCRIPTION:
RCT n = 50

Groups:

1. bridging
2. SCR

Outcomes:

1. WORC
2. ASES
3. QuickDASH
4. MRI at 12 months post-op

ELIGIBILITY:
Inclusion Criteria:

1. Large to massive rotator cuff tear (with or without subscapularis tear) that may possibly be irreparable without the use of graft materials (confirmed intra-operatively)
2. Either primary tear or re-tear after previous repair
3. Radiographic evidence of Hamada stage 1-3, with or without Samilson & Prieto mild osteoarthritis (<3mm inferior osteophyte)

Exclusion Criteria:

1. Primary glenohumeral osteoarthritis: radiographic evidence of Samilson & Prieto classification moderate or greater
2. Cuff tear arthropathy (CTA): radiographic evidence of Hamada stage 4 or above
3. Inflammatory joint disease of the shoulder (e.g. rheumatoid arthritis)
4. Medical issues precluding surgery
5. Unwilling or unable to complete study outcomes
6. Worker's Compensation Claim or litigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2020-11-07 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
American Shoulder and Elbow Surgeon Outcome - patient portion | 24 months
  American Shoulder and Elbow Surgeon Outcome - patient portion (minimum score = 0, maximum score = 100, best outcome = 100)
American Shoulder and Elbow Surgeon Outcome - patient portion | 12 months
  American Shoulder and Elbow Surgeon Outcome - patient portion (minimum score = 0, maximum score = 100, best outcome = 100)
American Shoulder and Elbow Surgeon Outcome - patient portion | 6 months
  American Shoulder and Elbow Surgeon Outcome - patient portion (minimum score = 0, maximum score = 100, best outcome = 100)
American Shoulder and Elbow Surgeon Outcome - patient portion | 3 months
  American Shoulder and Elbow Surgeon Outcome - patient portion (minimum score = 0, maximum score = 100, best outcome = 100)

SECONDARY OUTCOMES:
Western Ontario Rotator Cuff Index | 24 months
  Western Ontario Rotator Cuff Index (score converted to /100, minimum = 0, maximum = 100, best outcome = 100)
Western Ontario Rotator Cuff Index | 12 months
  Western Ontario Rotator Cuff Index (score converted to /100, minimum = 0, maximum = 100, best outcome = 100)
Western Ontario Rotator Cuff Index | 6 months
  Western Ontario Rotator Cuff Index (score converted to /100, minimum = 0, maximum = 100, best outcome = 100)
Western Ontario Rotator Cuff Index | 3 months
  Western Ontario Rotator Cuff Index (score converted to /100, minimum = 0, maximum = 100, best outcome = 100)
Disabilities of the Arm, Shoulder and Hand - QuickDASH | 24 months
  Disabilities of the Arm, Shoulder and Hand - QuickDASH (minimum = 100, maximum = 0, best outcome = 0)
Disabilities of the Arm, Shoulder and Hand - QuickDASH | 12 months
  Disabilities of the Arm, Shoulder and Hand - QuickDASH (minimum = 100, maximum = 0, best outcome = 0)
Disabilities of the Arm, Shoulder and Hand - QuickDASH | 6 months
  Disabilities of the Arm, Shoulder and Hand - QuickDASH (minimum = 100, maximum = 0, best outcome = 0)
Disabilities of the Arm, Shoulder and Hand - QuickDASH | 3 months
  Disabilities of the Arm, Shoulder and Hand - QuickDASH (minimum = 100, maximum = 0, best outcome = 0)
Tendon healing, assessed via MRI | 12 months
  Tendon healing (classifications: intact or retorn)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Lo, MD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data.